CLINICAL TRIAL: NCT00002020
Title: Trial of an Alternative Dosing Regimen of Oral Retrovir in Patients With AIDS or Advanced ARC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Glaxo Wellcome (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 014L; 28
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1992-02

CONDITIONS: HIV Infections
Keywords: Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Zidovudine
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Zidovudine

INTERVENTIONS:
Drug: Zidovudine

SUMMARY:
To evaluate the safety and tolerance, in patients with severe clinical manifestations of HIV infection, of zidovudine (AZT) administered daily for 48 weeks as a low dose every 4 hours or a higher dose every 12 hours.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

- Prophylaxis or treatment for Pneumocystis carinii pneumonia (PCP) consisting of either trimethoprim / sulfamethoxazole, aerosolized pentamidine, pyrimethamine / sulfadoxine, or dapsone allowed at the discretion of the investigator.

Patients with the following are excluded:

* Any immediately life-threatening infection or medical condition present at the time of study entry.
* Any active opportunistic or other infection requiring chronic therapy at the time of study entry. Patients with PCP may be randomized to study medication following a minimum 7-day course of therapy resulting in stabilization of their disease. Patients with stabilized disease must have a fever < 39 C for at least 48 hours, pO2 (on room air ) = or > 60 mm, and an Arterial/alveolar gradient = or < 30 mm.
* Diagnosis of AIDS Dementia Complex.
* Received more than 4 weeks of antiretroviral therapy or who previously discontinued antiretroviral therapy due to drug related toxicity.
* Diseases and conditions listed in Exclusion Co-existing Conditions.

Patients must have the following:

* Seropositive for HIV infection documented by any federally licensed ELISA and confirmed by Western blot.
* Advanced HIV disease or AIDS-related complex.
* Ability to give informed consent.

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions or symptoms are excluded:

* AIDS with malignant disease likely to require cytotoxic chemotherapy.
* Diagnosis of AIDS Dementia Complex.
* Impaired renal function ( Creatinine clearance < 50 ml/min/1.73m2 or serum creatinine = or > 2 mg/dl).
* Impaired hepatic function ( ALT = or > 5 x upper limit of normal).
* Fever > 39 C at entry.

Concurrent Medication:

Excluded:

* Any other experimental therapy.
* Drugs which cause significant bone marrow suppression.
* Cytolytic chemotherapy.
* Drugs which cause significant nephrotoxicity or hepatotoxicity.

Concurrent Treatment:

Excluded:

* Radiation therapy (with the exception of electron beam therapy to an area < 100 cm2).

Prior Medication:

Excluded within 2 weeks of study entry:

- Any other experimental therapy. Drugs which cause significant bone marrow suppression. Cytolytic chemotherapy. Drugs which cause significant nephrotoxicity or hepatotoxicity.

Excluded within 4 weeks of entry:

- Immunomodulating agents, including pharmacological doses of steroids for more than 10 days (except for management of severe PCP in which case duration should not exceed 21 days). Interferon. Isoprinosine. IL-2.

Excluded within 8 weeks of entry:

-

Antiretroviral agents including:

- Ribavirin. Dideoxycytidine (ddC). Dideoxyadenosine (ddA). Didanosine (ddI). Foscarnet. Dextran Sulfate. AL-721. Retrovir (Zidovudine, AZT) for greater than 4 weeks or within 90 days of study entry, or patients who originally discontinued Retrovir due to drug-related toxicity. Drugs metabolized by hepatic glucuronidation may alter the metabolism of Retrovir and should not be used chronically.

Prior Treatment:

Excluded:

* Radiation therapy (with the exception of electron beam therapy to an area < 100 cm2) within 2 weeks of study entry.

Known active drug or alcohol abuse.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (12):
- United States (11):
  - Univ of Arizona / Health Science Ctr, Tucson, Arizona
  - Northwestern Univ Med School, Chicago, Illinois
  - Cook County Hosp, Chicago, Illinois
  - Rush Presbyterian - Saint Luke's Med Ctr, Chicago, Illinois
  - Univ of Missouri at Kansas City School of Medicine, Kansas City, Missouri
  - North Jersey Community Research Initiative, Newark, New Jersey
  - Univ of New Mexico Hlth Sciences Ctr / Dept of Med, Albuquerque, New Mexico
  - Northshore Hosp / Cornell Univ, Manhasset, New York
  - Univ of Pennsylvania / HIV Clinic, Philadelphia, Pennsylvania
  - Univ TX Galveston Med Branch, Galveston, Texas
  - Baylor College of Medicine, Houston, Texas
- San Juan Veterans Administration Med Ctr, San Juan, Puerto Rico